CLINICAL TRIAL: NCT05289843
Title: Effect of Rosmarinus Officinalis Versus 2.5%Sodium Hypochlorite as Root Canal Irrigants on the Intensity of Post-operative Pain and Bacterial Reduction in Asymptomatic Necrotic Mandibular Premolars
Brief Title: Rosmarinus Officinalis Versus 2.5%Sodium Hypochlorite as Root Canal Irrigants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayah Tarek El Sayed Abudlaah, Principal investigator and Master degree student at faculty of dentistry , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO 3-7-2
Record Dates: First submitted 2022-02-09; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant , Investigator, Outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Rosmarinus officinals will be used as root canal irrigant in treating aysymptomatic mandibular premolars.
  Interventions: Other: Rosmarinus Officinallis
- Control Group (No Intervention): Sodium Hypochlorite used as control in root canal irrigations in treating a asymptomatic mandibular premoalrs.

INTERVENTIONS:
Other: Rosmarinus Officinallis — Root canal Irrigants
  Arms: Experimental

SUMMARY:
To measure the Effect of Rosmarinus Officinalis versus 2.5%Sodium Hypochlorite as Root canal Irrigants on the Intensity of post-operative pain and Bacterial Reduction in asymptomatic necrotic Mandibular premolars.

ELIGIBILITY:
Inclusion Criteria:

1. Systematically healthy patient (ASA I and II).
2. Age between 20 and 45 years with no sex predilection
3. Mandibular permanent premolar teeth:

   * Diagnosed clinically with pulp necrosis.
   * Absence of spontaneous pain.
   * Radiographic evidence of root and root canal.
   * Slight widening in the periodontal membrane space or with periapical radiolucency.
   * No response to cold pulp tester (ethyl chloride spray)
4. Patients who can understand and interpret Numerical rating scale (NRS).
5. Patients' acceptance to participate in the trial

Exclusion Criteria:

* 1- Medically compromised patients having significant systemic disorders. (ASA III or IV).

  2- History of intolerance to NSAIDS. 3- If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively as it might alter their pain perception.

  4- Pregnant women: Avoid radiation exposure, anesthesia, and medication. 5- Teeth with: i. Vital teeth. ii. Double canal mandibular premolar teeth iii. Association with swelling or fistulous tract. iv. Acute peri-apical abscess and swelling: Need special treatment steps which could involve additional visits with incision and drainage. Also, it could influence initiation and progression of postoperative pain.

  v. Mobility Grade II or III. vi. Pocket depth more than 5mm. vii. Previous root canal therapy. viii. Non-restorable teeth: Hopeless tooth
* Immature teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain after root canal treatment. | Up to 48 hours postoperative.
  The patient is asked to grade his degree of pain on the Numerical Rating Scale (NRS) chart which is an 11 points scale consisting of numbers from 0 to 10, where zero reading represents no pain , 1-3 readings represent mild pain, 4-6 readings represent moderate pain. 7-10 readings represent severe pain .

SECONDARY OUTCOMES:
Intracanal bacterial load change. | First as a base line and after 15 minutes ( End of the chemo-mechanical preparation).
  The intracanal bacterial load change is calculated through using colony forming units per milliliter test before and after root canal preparation.